CLINICAL TRIAL: NCT00102388
Title: Efficacy and Safety of Vildagliptin Compared to Gliclazide in Drug Naive Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLAF237A2310
Record Dates: First submitted 2005-01-29; First posted 2005-01-31 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: type 2 diabetes; vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; Gliclazide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- vildagliptin (Experimental)
  Interventions: Drug: vildagliptin
- Gliclazide (Active Comparator)
  Interventions: Drug: Gliclazide

INTERVENTIONS:
Drug: vildagliptin
  Arms: vildagliptin
Drug: Gliclazide
  Arms: Gliclazide

SUMMARY:
This study is not being conducted in the United States. The purpose of this study is to assess the safety and effectiveness of vildagliptin, an unapproved drug, compared to gliclazide in lowering overall blood glucose levels in people with type 2 diabetes who have not been previously treated with drug therapy to lower their blood sugar.

ELIGIBILITY:
Inclusion Criteria:

* Not currently on drug therapy for type 2 diabetes
* Body mass index (BMI) in the range 22-45
* Blood glucose criteria must be met

Exclusion Criteria:

* Pregnancy or lactation
* Type 1 diabetes
* Evidence of significant diabetic complications
* Evidence of serious cardiovascular conditions
* Laboratory value abnormalities as defined by the protocol
* Other protocol-defined exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1092 (Actual)
Dates: Start 2005-01; Primary Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c at 104 weeks | 104 weeks

SECONDARY OUTCOMES:
Adverse event profile at 104 weeks | 104 weeks
Change from baseline in fasting plasma glucose at 104 weeks | 104 weeks
Patients with endpoint HbA1c <7% after 104 weeks | 104 weeks
Patients with reduction in HbA1c >/= 0.7% after 104 weeks | 104 weeks
Patients with reduction in HbA1x >/= 0.5% after 104 weeks | 104 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Investigative Site, Investigative Centers, Germany
- Novartis Pharmaceuticals, Basel, Switzerland

REFERENCES:
- [Result] Foley JE, Sreenan S. Efficacy and safety comparison between the DPP-4 inhibitor vildagliptin and the sulfonylurea gliclazide after two years of monotherapy in drug-naive patients with type 2 diabetes. Horm Metab Res. 2009 Dec;41(12):905-9. doi: 10.1055/s-0029-1234042. Epub 2009 Aug 24. PMID 19705345
- [Result] Filozof C, Schwartz S, Foley JE. Effect of vildagliptin as add-on therapy to a low-dose metformin. World J Diabetes. 2010 Mar 15;1(1):19-26. doi: 10.4239/wjd.v1.i1.19. PMID 21537424
- [Result] Goodman M, Thurston H, Penman J. Efficacy and tolerability of vildagliptin in patients with type 2 diabetes inadequately controlled with metformin monotherapy. Horm Metab Res. 2009 May;41(5):368-73. doi: 10.1055/s-0028-1104604. Epub 2009 Feb 16. PMID 19221978